CLINICAL TRIAL: NCT00705211
Title: Designated Drug Use Investigation (Long-Term Administration) of Zetia 10-mg Tablets - A 52-Week Long-Term Designated Drug Use Investigation of Zetia Monotherapy and Combination Therapy
Brief Title: A 52-week Post-marketing, Observational Study to Confirm the Safety and Efficacy of Zetia Alone or in Combination With Other Lipid-lowering Drugs in Japanese Subjects With Hypercholesterolemia (Study P05245)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: P05245
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Familial Hypercholesterolemia; Homozygous Sitosterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Zetia monotherapy: Patients to be treated with Zetia alone (10-mg tablets,) for hypercholesterolemia
  Interventions: Drug: Ezetimibe
- Zetia combination therapy: Patients to be treated with Zetia (10-mg tablets,) in combination with other lipid-lowering drugs for hypercholesterolemia
  Interventions: Drug: Ezetimibe + other lipid-lowering medication(s)

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe, 10-mg tablets,
  Other Names: Zetia
  Groups: Zetia monotherapy
Drug: Ezetimibe + other lipid-lowering medication(s) — Ezetimibe, 10-mg tablets, other lipid-lowering medication(s) as prescribed by attending physician
  Other Names: Zetia + other lipid-lowering medication(s)
  Groups: Zetia combination therapy

SUMMARY:
This study is a non-interventional (observational) study in Japan to confirm the safety and efficacy of Zetia when administered alone or in combination with other lipid-lowering drugs in daily medical practice throughout a 52-week period. It is being conducted as a post-approval commitment, in accordance with the Ministry of Health, Labour and Welfare's guideline on Good Post-marketing Study Practice.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

DETAILED DESCRIPTION:
The population will be selected from 200 institutions in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have hypercholesterolemia, familial hypercholesterolemia, or homozygous sitosterolemia will be considered for this study.

Zetia monotherapy patients must be treated with Zetia alone.

Zetia combination therapy patients must be treated with Zetia in combination with other lipid-lowering drugs for hypercholesterolemia.

Exclusion Criteria:

* Patients with a history of hypersensitivity to any ingredient in Zetia
* Patients with serious hepatic function disorder should not be treated with Zetia in combination with an HMG-CoA reductase inhibitor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population will be selected from 200 institutions in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 1794 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
A primary endpoint is the incidence of adverse events. | Adverse events will be monitored throughout the 52-week period. (Subjects who discontinue Zetia treatment during the 52-week period will be investigated up to the time of therapy discontinuation.)
A primary endpoint is change in LDL-C | LDL-C at start of 52 weeks will be compared to LDL-C at the end of the 52-week period. (Subjects who discontinue Zetia treatment during the 52-week period will be investigated up to the time of therapy discontinuation.)